CLINICAL TRIAL: NCT07182851
Title: Prevalence of Pain in Mechanically Ventilated Patients in Intensive Care Units
Acronym: PainICU
Status: Recruiting | Type: Observational
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Hospital Central da Aeronáutica, Rio de Janeiro (Unknown); Hospital Universitário Clementino Fraga Filho (Other); Hospital Universitário Gafrée Guinle (Unknown); Hospital Central da Polícia Militar do Estado do Rio de Janeiro (Unknown); Hospital Doutor João Felício (Unknown)
Responsible Party: Sponsor
Other Study IDs: pain_icu_unisuam_2025
Record Dates: First submitted 2025-06-03; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Sedation and Analgesia; Pain Intensity Assessment; Mechanical Ventilation Complication
Keywords: mechanical ventilation; intensive care unit; Pain Assessment
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Pain is a subjective symptom, a physiological response that is difficult to assess, which affects the body physically and/or emotionally. It is a common phenomenon among clinical and surgical patients in Intensive Care Units (ICU). And its effects are the combined results of physiological and behavioral aggressions caused by clinical conditions, immobility and the execution of common procedures in ICU's. The presence of pain appears to be independently associated with worse clinical outcomes, including higher infection rates, patient-ventilator asynchronies, delirium, prolonged mechanical ventilation (MV), length of hospital stay and higher healthcare costs. Objectives: To evaluate the prevalence of pain and its associated factors in mechanically ventilated surgical patients in ICU's. Methods: This is a cohort, prospective, multicenter study designed to estimate the prevalence of pain, its intensity, its associated factors, correlating them to outcomes such as patient-ventilator asynchrony rate, time to weaning, and 28-day mortality in mechanically ventilated patients. All research participants who meet the inclusion criteria and who are not using neuromuscular blockers, or have any other condition associated with altered pain perception, will be evaluated using the Behavioral Pain Scale (BPS) and the Critical Care Pain Observation Tool (CPOT) on the 2nd day of mechanical ventilation and on the first day of awakening, when the RASS scale is between 4 and -2. At the same time, data will be collected on the ongoing sedoanalegesia strategy, and the asynchrony index will be calculated [(Nº of asynchronous ventilatory cycles/Nº of ventilatory cycles studied) *100]. The end point of the research will be 28 days, where the time until weaning, time until discharge or death will be established using the Kaplan-Meier estimators. Expected results: The prevalence of pain and its intensity is associated with the presence of patient-ventilator asynchronies and thus with harsh outcomes related to the length of stay in the ICU, time until weaning and thirty-day mortality in the ICU. It is estimated that there is agreement between the BPS and CPOT scales in mechanically ventilated patients.

DETAILED DESCRIPTION:
PARTICIPANTS AND METHODS

ETHICAL ASPECTS

This project was submitted to the Ethics and Research Committee (CEP) of UNISUAM, via Platform Brazil, by the project coordinating center and will have the consent of all participating institutions, as per and predicted in the standards from the Resolution 466/12, of Advice National of Health (CNS) (Brazil, 2012) and in Law 14,874/2024, which establishes the National System of Ethics in Research with Human Beings (Brazil, 2024) and approved under number: 83431424.8.1001.5235 . Like this, the investigators ensure what principles ethical will be followed to the far away from the search, with one commitment explicit of respect the autonomy and these values of participants, while ensuring the confidentiality of data. All data will be reported later following the recommendations of STROBE ( STRengthening the Reporting of Observational studies in Epidemiology).

LOCATION OF REALIZATION OF STUDY

The study will be a multicenter study involving public and private hospitals, with the coordinating center of the study being the Augusto Motta University Center

SAMPLE

The sample size for qualitative variable and quantity variables are different and were based on previously study . Thus, as our primary outcome will be the assessment of the prevalence of pain in mechanically ventilated patients and this classification will be dichotomous, the investigators will use the sample calculation for qualitative variables.

For qualitative variable

To find out the proportion of patients who experience considerable pain in the ICU (BPS > or = 5) in a population, the investigators use the formula below since this proportion is qualitative.

Sample size = [ Z 1-α/2 2 xpx(1-p)]/d 2 ]

Being:

Z 1-α/2 = It is a standard normal variable (assuming 5% type 1 error (p<0.05) it is 1.96 and with 1% type 1 error (P<0.01) it would be 2.58). Since in most studies P values are considered significant below 0.05, therefore 1.96 was used in the formula.

p = Expected proportion in the population based on previous studies d = Absolute error or precision - sênior investigators decided on an absolute error of 5%

In this case, to estimate the proportion of participants with considerable pain experience (BPS ≥ 5) in volunteers admitted to intensive care units under mechanical ventilation and in accordance with previous studies that establish an estimate of a BPS ≥ 5 at 40%, the sample size was calculated with a precision error of 5% and a type 1 error percentage of 5%.

Sample size = [1.96 2 x 0.4 x(1-0.4)]/0.05 2

Therefore, for this cohort, multicenter study, 370 participants will be evaluated .

LOCATION OF RECRUITMENT

All participants will be recruited from the ICUs of participating hospitals between june and december to 2025.

PROCEDURES

STANDARDIZATION OF COLLECTION PROCEDURES

Researchers from the study's Coordinating Center will conduct online training with the heads of each participating center and will provide an instructional video on the collection procedures. All data will be entered into a database with input masking and coded using Research Electronic Data Capture (REDCap).

CLINICAL DATA

Data on age, sex, body weight, height, surgery, SAPS 3 score ( Simplified Acute Physiology Score 3) and Sequential Organ Failure Assessment (SOFA) will be collected at the time of ICU admission. Information on time to successful weaning from mechanical ventilation, time to successful discharge from the ICU and 28-day hospital mortality will also be collected.

PROCEDURES

All participants will be evaluated at two moments: second day after mechanical ventilation and on the first day of sedation suspension, with superficialization confirmed by a RASS ≤ -2 (-2 to +2). The evaluations will always occur at the same time, in the morning, after the routine tracheal aspiration procedure (which is known to be one of the main causes of pain in mechanically ventilated patients). All evaluation procedures will occur during the first physiotherapy appointment during the daytime period on the respective days.

Pain will be assessed by the Behavioral Pain Scale and the Critical Care Pain Observation Tool, which are tools validated in Brazil and are widely used to assess critically ill, uncooperative patients.

At this time, the asynchrony index (AI, %) will also be evaluated, calculated as the ratio between the number of asynchronous cycles/total ventilatory cycles studied X 100.

These assessments will be carried out at least 1 hour after bathing or nursing care procedures to wash out any painful experiences that may arise.

The entire pharmacological strategy will be expressed in dose/weight/time. Patients will be divided into two groups: a "pain" group in which BPS ≥ 5 and a "no pain" group in which BPS < 5. The criterion for establishing the cutoff point at BPS values BPS ≥ 5 was determined based on previous studies that defined it as a "pain event", or as an "inadequate state" of pain.

ANALYSIS OF DATA

The data will be collected by the coordinators or routines of the ICUs of the participating centers, using an input mask, being coded and later evaluated by an independent statistician, who did not participate or will not participate in any stage of the project execution.

FLAT OF ANALYSIS STATISTIC

Results will be expressed as numbers (%) for categorical variables and medians (interquartile range) for continuous variables. The primary outcome measure for this project will be pain intensity before and after a painful stimulation procedure using the BPS on a scale of 3 to 12 and the CPOT on a scale of 0 to 8.

Univariate logistic regression analysis will be used to identify parameters associated with pain events in the event group. Normality of data will be checked using the Kolmogorov-Smirnov test, while homogeneity of variance will be checked by the F test. Student's t-test or Welch's test, or the Wilcoxon test will be used for continuous data, as appropriate. Chi-square or Fisher's exact test will be used for categorical variables. After that, a multivariate logistic regression analysis will be used to determine factors independently associated with pain in the groups categorized as "pain" (BPS ≥ 5) or "no pain" (BPS < 5). Variables will be entered into a model when they were associated with pain status.

This will be based on a univariate logistic regression analysis significance threshold of p < 0.1, and when there is no mutual correlation, based on a Spearman correlation coefficient greater than 0.7 or less than -0.7. The final model will be constructed using backward elimination of non-significant variables. Odds ratios and 95% confidence intervals (95% CI) will be calculated based on the likelihood ratio statistic. Comparative analyses of the three components of the BPS and CPOT will be performed using the Friedman test followed by the Dunn test and multiple comparison test. Univariate analysis of clinical outcomes will be performed for time to successful weaning from mechanical ventilation, time to ICU discharge, as well as 30-day in-hospital mortality rate using the log-rank test. In addition to these univariate analyses, clinical outcomes will be assessed using multivariate analyses.

Logistic regression analysis, correcting for risk factors, will use variables that present at least a trend towards significance (p < 0.1) in the univariate analysis. The parameters will be checked for linearity and non-linear parameters will be entered into the model as nominal variables. Odds ratios as well as 95% CI will be calculated for the outcomes. All values that result in two-sided statistical tests with a p value ≤ 0.05 will be considered significant. R statistics (R, version 2.15.2) were used to analyze the data. The analyses will be computed using R Software (version 2.15.2).

AVAILABILITY OF ACCESS TO THE DATA

All data of present study will be available through of one universal data repository, in addition to the virtual library and database of UNISUAM and each center participating in the study

RESULTS EXPECTED

This research project will provide a current data set on pain in mechanically ventilated patients, using two validated tools for this screening and will correlate the presence of pain with clinical factors, sedation and analgesia regimen employed, with the presence of patient-ventilator asynchrony and thus with hard outcomes related to length of stay in the ICU, time to weaning and 28-day mortality in the ICU.

ELIGIBILITY:
Inclusion Criteria

Participants of both sexes, aged 18 or over;

Participants who are using invasive mechanical ventilation,

Exclusion Criteria:

Participants undergoing treatment with neuromuscular blockers,;

Participants with any condition associated with altered pain perception (e.g., Guillain-Barré Syndrome, SCI, etc.);

Participants with any condition that would likely interfere with behavioral assessments of pain (e.g., decortication or decerebration posture)

As the assessments will be carried out before and after the tracheal aspiration procedure, if the patient does not have objective criteria for tracheal aspiration, he/she will be excluded from the study, irrefutably preventing the procedure from being carried out without express need.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patientes admitted in ICU's in use of invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity by BPS | From second day after enrollment , from first day at RASS -2 or minus, with end point 28 - day.
  The intensity of pain will be assessment by Behavioral Pain Scale (BPS) in the morning, after the first tracheal suctioning procedure.
Pain intensity by CPOT | Time Frame: From second day after enrollment , from first day at RASS -2 or minus, with end point 28 - day.
  The intensity of pain will be assessment by Critical care pain observation tool (CPOT) in the morning after the first tracheal suctioning procedure.

SECONDARY OUTCOMES:
Ventilatory Settings | From second day after enrollment, from first day at RASS-2 or minus, with end point 28-day"
  All participants will be evaluated in relation to the ventilatory parameters used in the pain assessment measurement.
Airway occlusion pressure(P0.1) | This measurement will be taken on the second day of mechanical ventilation and on the first day after reduction or suspension of sedation in which the patient assumes a RASS -2 or less. The study endpoint will be in 28 days.
  All participants will have their expiratory occlusion pressure measured in the first 100 milliseconds of inspiration(P0.1, cmH2O), using the mechanical ventilator's own algorithm. When the P0.1 measurement button is pressed, the inspiratory flow valve is closed to prevent gas from flowing into the lungs during the measurement.
  The pressure is recorded 100 ms after the start of the inspiratory effort. Three measurements will be taken with a 1-minute interval between each one. The average of the three measurements will be calculated according to previous studies.
Patient-mechanical ventilator asynchrony index | This asynchrony index will be measured on the second day of mechanical ventilation and on the first day after suspension or reduction of sedation with the participant assuming a RASS-2 or less. The study endpoint will be 28 days.
  The asynchrony index (AI) was defined by previous studies by the number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (patient-triggered) and of wasted efforts: asynchrony index (expressed in percentage) = number of asynchrony events/total respiratory rate (ventilator cycles + ineffective triggering) × 100. As previously reported, a high incidence of asynchrony was defined as an asynchrony index greater than 10%.
28-day mortality | 28 days
  Proportion of participants who died within 28 days after randomization/study enrollment
Duration of mechanical ventilation | Up to 28 days or hospital discharge, whichever occurs first
  Total time (in days or hours) on invasive mechanical ventilation from initiation to definitive discontinuation or death
Time to weaning from mechanical ventilation | Up to 28 days
  Time (in days or hours) from initiation of mechanical ventilation to successful weaning (defined as discontinuation of mechanical ventilation for at least 48 consecutive hours without need for reintubation)

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Hospital Central da Aeronáutica, Rio de Janeiro, Rio de Janeiro
  - Hospital Central da Polícia Militar do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Gafrée Guinle, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Yes
You data of present study will be available through of one universal data repository, in addition to the virtual library and database of UNISUAM and each center participating in the study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From december 2025 for 5 five years